CLINICAL TRIAL: NCT04029532
Title: Factors Associated With Obesity in Adult Women: Respiratory Exchange Ratio, Heart Rate Variation and Body Image
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201901140RINA
Record Dates: First submitted 2019-04-15; First posted 2019-07-23 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2019-11

CONDITIONS: Obesity
Keywords: Respiratory exchange ratio; Body image; Heart rate variability
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-overweight/obese & normal weight: Body mass index (BMI) < 24.0 kg/m^2
  Interventions: Device: Respiratory exchange ratio; Device: Heart rate variability; Device: Body composition; Behavioral: Eating behavior; Behavioral: Physical activity recall; Behavioral: Depression; Behavioral: Body image
- Overweight and obese: Body mass index (BMI) >= 24.0 kg/m^2
  Interventions: Device: Respiratory exchange ratio; Device: Heart rate variability; Device: Body composition; Behavioral: Eating behavior; Behavioral: Physical activity recall; Behavioral: Depression; Behavioral: Body image

INTERVENTIONS:
Device: Respiratory exchange ratio — Ask participants to supine on bed, using a ventilator hood cover upon their head. Measure respiratory exchange ratio for 15 minutes.
Device: Heart rate variability — Ask participants to supine on bed for 10 minutes, connect electrodes on their right wrist. Measure heart rate variability for 5 minutes.
Device: Body composition — Ask participants to supine on bed for 10 minutes, connect electrodes on their right wrist and right foot. Measure body composition.
Behavioral: Eating behavior — Fill in questionnaire (Three-Factor Eating Questionnaire, revised 18-item, TFEQ-18).
Behavioral: Physical activity recall — Fill in questionnaire (Seven-days Physical Activity Recall, 7-d PAR).
Behavioral: Depression — Fill in questionnaire (Mongomery-Asberg Depression Rating Scale, MADRS).
Behavioral: Body image — Fill in questionnaire (multi-directional self-body relationship questionnaire (MBSRQ), figure rating scale (FRS)).

SUMMARY:
The prevalence of obesity all over the world has increased year by year, and how to effectively prevent and treat obesity has become an important health care issue. Many adjustable and nonadjustable causes of obesity have been proposed, such as unbalanced eating habits, lack of physical activity, psychological factors, and genes. The practice guidelines recommended lifestyle modification interventions which include diet control combined with regular exercise as the core treatment for obesity, but the effects on different ethnic groups are not ideal. In order to provide more choices for future weight loss intervention, it would be important to find out more risk factors for obesity. Previous studies have shown that lower sympathetic activity assessed by heart rate variability was related to obesity; obese men have higher respiratory exchange rates which might indicate they are more likely to use carbohydrates as a source of energy, and therefore, fat cannot be effectively consumed and led to an accumulation in the body. Furthermore, previous studies showed that Asians are less satisfied with their body image than other races, and women are more dissatisfied than men. Poor body image will lead to a series of effects, such as changes in eating habits, hormonal changes, depression, etc., eventually forming a vicious circle of obesity. However, most aforementioned Asians in these studies are immigrants living in overseas areas such as the Americas, and cannot fully represent the ethnic groups in Asia. Therefore, the purpose of this study are (1) to investigate the physiological and psychological factors influence obesity in adult women, including respiratory exchange rate, heart rate variability, and body image, and (2) to examine the correlations among these risk factors and different degree of obesity.

DETAILED DESCRIPTION:
Methods: This is a cross-sectional design study. Subjects were recruited from Taipei city. Inclusion criteria are women aged between 20 and 50 years old and have willing to participate to this study. Subjects will be excluded as follows: (1) taking medications that affect weight or hormones; (2) fluctuation of weight exceeds 2 kg within 3 months before the enrolled in study; (3) any condition that causes the subject fail to complete the test paper, such as: cognitive problems; (4) diagnosed with mental illness; (5) pregnancy or menopause. The assessments include: obesity-related indicators (height, weight, waist and hip circumference, percentage of body fat), respiratory exchange ratio, heart rate variability, body image (multi-directional self-body relationship questionnaire (MBSRQ), figure rating scale (FRS)), physical activity (Seven-days Physical Activity Recall, 7-d PAR), eating behavior (Three-Factor Eating Questionnaire, revised 18-item, TFEQ-18), and depression (Mongomery-Asberg Depression Rating Scale, MADRS). Statistical analysis will be performed by using SPSS version 18 (SPSS Inc, Chicago: SPSS Inc.), and significant level would be set at 0.05. Analysis of variance (ANOVA) will be used to examine the differences of all measured variables among different degrees of obesity groups. In addition, we will use multiple linear regression analysis to examine whether overweight and obesity are significantly related to respiratory exchange rate, heart rate variability and body image.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years old, premenopausal

Exclusion Criteria:

* Taking medications that affect weight or hormones
* Fluctuation of weight exceeds 2 kg within 3 months before the enrolled in study
* Any condition that causes the subject fail to complete the test paper, such as: cognitive problems
* Diagnosed with mental illness
* Pregnancy or menopause

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenopausal women
Study Population: Asian, mainly living in Taiwan
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-26 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Respiratory exchange ratio (RER) | After filling in all questionnaires, lasting 15 minutes.
  Ask participants to supine on bed, using a ventilator hood cover upon their head. Measure respiratory exchange ratio for 15 minutes.
  Device used: Vmax® Encore Metabolic Cart, Carefusion Corporation, Yorba Linda, California (CA).
  Normal range: 0.7-1.0, greater value indicates more carbohydrates oxidation, while smaller value indicates more fat oxidation.
Heart rate variability (HRV) | After measuring respiratory exchange ratio, lasting 15 minutes.
  Ask participants to supine on bed for 10 minutes, connect electrodes on their right wrist. Measure heart rate variability for 5 minutes. Device used: SS1C, Enjoy Research Inc., Taiwan.
  High frequency (HF): greater value indicates active parasympathetic activity. Low frequency-high frequency ratio (LF/HF): greater value indicates active sympathetic activity.
Body image | After filling in basic data questionnaire, lasting 10 minutes.
  Fill in questionnaire (multi-directional self-body relationship questionnaire (MBSRQ)). There are 69 questions, each question scores 1-5 points. Sum up all points, greater value indicates better body image.
Body image (evaluative component) | After filling in multi-directional self-body relationship questionnaire (MBSRQ), lasting 5 minutes.
  Figure rating scale (FRS) is used. Nine figures of women (from lean to obese) is provided, participants are asked to choose which figure fits her present and ideal appearance the most. Scoring 1-9 points, greater value indicates poorer body image.

SECONDARY OUTCOMES:
Body fat percentage | After measuring heart rate variability, lasting 5 minutes.
  Ask participants to supine on bed for 10 minutes, connect electrodes on their right wrist and right foot. Measure body fat percentage. Device used: Maltron BioScan 920-2. Greater value indicates higher body fat percentage.
Physical activity | After filling in body image questionnaire, lasting 5 minutes.
  Fill in questionnaire (Seven-days Physical Activity Recall, 7-d PAR). Participants are asked to recall average time spent in a week on sleeping and activities of different intensities (Unit: metabolic equivalent of tasks (METs)). Sleeping, mild activity, moderate activity, vigorous activity, very vigorous activity are calculated as 1, 1.5, 4, 6, 10 METs respectively. Sum up all METs, divided by 7, we can obtain average daily energy expenditure. Greater value indicates more physical activity done.
Eating behavior | After filling in physical activity questionnaire, lasting 5 minutes.
  Fill in questionnaire (Three-Factor Eating Questionnaire, revised 18-item, TFEQ-18). This questionnaire includes 18 questions, scoring 1-4 points, except question 18 (1-8 points). Sum up all points, greater value indicates better eating behavior.
Depression | After filling in eating behavior questionnaire, lasting 5 minutes.
  Fill in questionnaire (Mongomery-Asberg Depression Rating Scale, MADRS). This questionnaire includes 10 questions, scoring 0-6 points. Sum up all points, greater value indicates more depressed.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, College of Medicine, Department of Physical Therapy, Taipei, Zhongzheng, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We will respect the participants' willingness.

REFERENCES:
- [Background] Hruby A, Hu FB. The Epidemiology of Obesity: A Big Picture. Pharmacoeconomics. 2015 Jul;33(7):673-89. doi: 10.1007/s40273-014-0243-x. PMID 25471927
- [Background] Acosta A, Streett S, Kroh MD, Cheskin LJ, Saunders KH, Kurian M, Schofield M, Barlow SE, Aronne L. White Paper AGA: POWER - Practice Guide on Obesity and Weight Management, Education, and Resources. Clin Gastroenterol Hepatol. 2017 May;15(5):631-649.e10. doi: 10.1016/j.cgh.2016.10.023. Epub 2017 Feb 27. PMID 28242319
- [Background] Ryan DH, Kahan S. Guideline Recommendations for Obesity Management. Med Clin North Am. 2018 Jan;102(1):49-63. doi: 10.1016/j.mcna.2017.08.006. PMID 29156187
- [Background] Ramos-Jimenez A, Hernandez-Torres RP, Torres-Duran PV, Romero-Gonzalez J, Mascher D, Posadas-Romero C, Juarez-Oropeza MA. The Respiratory Exchange Ratio is Associated with Fitness Indicators Both in Trained and Untrained Men: A Possible Application for People with Reduced Exercise Tolerance. Clin Med Circ Respirat Pulm Med. 2008 Feb 1;2:1-9. doi: 10.4137/ccrpm.s449. PMID 21157516
- [Background] Weng KP, Ho TY, Ou SF, Lin CC, Hsieh KS. Heart rate variability analysis. Taiwan Medical Journal. 2009;52:290-3.
- [Background] Wang ML, Lin PL, Huang CH, Huang HH. Decreased Parasympathetic Activity of Heart Rate Variability During Anticipation of Night Duty in Anesthesiology Residents. Anesth Analg. 2018 Mar;126(3):1013-1018. doi: 10.1213/ANE.0000000000002439. PMID 29200073
- [Background] Messina G, De Luca V, Viggiano A, Ascione A, Iannaccone T, Chieffi S, Monda M. Autonomic nervous system in the control of energy balance and body weight: personal contributions. Neurol Res Int. 2013;2013:639280. doi: 10.1155/2013/639280. Epub 2013 Apr 11. PMID 23691314
- [Background] Tonhajzerova I, Javorka M, Trunkvalterova Z, Chroma O, Javorkova J, Lazarova Z, Ciljakova M, Javorka K. Cardio-respiratory interaction and autonomic dysfunction in obesity. J Physiol Pharmacol. 2008 Dec;59 Suppl 6:709-18. PMID 19218698
- [Background] Rodriguez-Colon SM, Bixler EO, Li X, Vgontzas AN, Liao D. Obesity is associated with impaired cardiac autonomic modulation in children. Int J Pediatr Obes. 2011 Apr;6(2):128-34. doi: 10.3109/17477166.2010.490265. Epub 2010 Oct 4. PMID 20919806
- [Background] Karason K, Molgaard H, Wikstrand J, Sjostrom L. Heart rate variability in obesity and the effect of weight loss. Am J Cardiol. 1999 Apr 15;83(8):1242-7. doi: 10.1016/s0002-9149(99)00066-1. PMID 10215292
- [Background] Yadav RL, Yadav PK, Yadav LK, Agrawal K, Sah SK, Islam MN. Association between obesity and heart rate variability indices: an intuition toward cardiac autonomic alteration - a risk of CVD. Diabetes Metab Syndr Obes. 2017 Feb 17;10:57-64. doi: 10.2147/DMSO.S123935. eCollection 2017. PMID 28255249
- [Background] Sudarsana U, Shrestha S, Kumar P. Comparative analysis of autonomic function tests in normotensive premenopausal and postmenopausal women. Int J Med Res Prof. 2017;3;234-9.
- [Background] Monda M, Messina G, Vicidomini C, Viggiano A, Mangoni C, De Luca B. Activity of autonomic nervous system is related to body weight in pre-menopausal, but not in post-menopausal women. Nutr Neurosci. 2006 Jun-Aug;9(3-4):141-5. doi: 10.1080/10284150600903552. PMID 17176636
- [Background] Cash TF, Morrow JA, Hrabosky JI, Perry AA. How has body image changed? A cross-sectional investigation of college women and men from 1983 to 2001. J Consult Clin Psychol. 2004 Dec;72(6):1081-1089. doi: 10.1037/0022-006X.72.6.1081. PMID 15612854
- [Background] Schwartz MB, Brownell KD. Obesity and body image. Body Image. 2004 Jan;1(1):43-56. doi: 10.1016/S1740-1445(03)00007-X. PMID 18089140
- [Background] Weinberger NA, Kersting A, Riedel-Heller SG, Luck-Sikorski C. Body Dissatisfaction in Individuals with Obesity Compared to Normal-Weight Individuals: A Systematic Review and Meta-Analysis. Obes Facts. 2016;9(6):424-441. doi: 10.1159/000454837. Epub 2016 Dec 24. PMID 28013298
- [Background] Scheffers M, van Duijn MAJ, Bosscher RJ, Wiersma D, Schoevers RA, van Busschbach JT. Psychometric properties of the Dresden Body Image Questionnaire: A multiple-group confirmatory factor analysis across sex and age in a Dutch non-clinical sample. PLoS One. 2017 Jul 26;12(7):e0181908. doi: 10.1371/journal.pone.0181908. eCollection 2017. PMID 28746387
- [Background] Nuttall FQ. Body Mass Index: Obesity, BMI, and Health: A Critical Review. Nutr Today. 2015 May;50(3):117-128. doi: 10.1097/NT.0000000000000092. Epub 2015 Apr 7. PMID 27340299
- [Background] Schmidt SL, Kealey EH, Horton TJ, VonKaenel S, Bessesen DH. The effects of short-term overfeeding on energy expenditure and nutrient oxidation in obesity-prone and obesity-resistant individuals. Int J Obes (Lond). 2013 Sep;37(9):1192-7. doi: 10.1038/ijo.2012.202. Epub 2012 Dec 11. PMID 23229737
- [Background] World Health Organization. Obesity and overweight. http://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight，2018/9/1
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- [Background] Frames CW, Soangra R, Lockhart TE, Lach J, Ha DS, Roberto KA, Lieberman A. Dynamical Properties of Postural Control in Obese Community-Dwelling Older Adults dagger. Sensors (Basel). 2018 May 24;18(6):1692. doi: 10.3390/s18061692. PMID 29794998
- [Background] Silvestris E, de Pergola G, Rosania R, Loverro G. Obesity as disruptor of the female fertility. Reprod Biol Endocrinol. 2018 Mar 9;16(1):22. doi: 10.1186/s12958-018-0336-z. PMID 29523133
- [Background] Ho CS, Lu Y, Ndukwe N, Chew MW, Shabbir A, So JB, Ho RC. Symptoms of Anxiety and Depression in Obese Singaporeans: a Preliminary Study. East Asian Arch Psychiatry. 2018 Mar;28(1):3-8. PMID 29576551
- [Background] Tian S, Xu Y, Dong H. The effect of metabolic health and obesity phenotypes on risk of hypertension: A nationwide population-based study using 5 representative definitions of metabolic health. Medicine (Baltimore). 2018 Sep;97(38):e12425. doi: 10.1097/MD.0000000000012425. PMID 30235720
- [Background] Jung JY, Park SK, Oh CM, Ryoo JH, Choi JM, Choi YJ. The risk of type 2 diabetes mellitus according to the categories of body mass index: the Korean Genome and Epidemiology Study (KoGES). Acta Diabetol. 2018 May;55(5):479-484. doi: 10.1007/s00592-018-1112-4. Epub 2018 Feb 17. PMID 29455425
- [Background] Lin Y, Wang Y, Wu Q, Jin H, Ma G, Liu H, Wang M, Zhang Z, Chu H. Association between obesity and bladder cancer recurrence: A meta-analysis. Clin Chim Acta. 2018 May;480:41-46. doi: 10.1016/j.cca.2018.01.039. Epub 2018 Feb 20. PMID 29408169
- [Background] Leung AWY, Chan RSM, Sea MMM, Woo J. An Overview of Factors Associated with Adherence to Lifestyle Modification Programs for Weight Management in Adults. Int J Environ Res Public Health. 2017 Aug 16;14(8):922. doi: 10.3390/ijerph14080922. PMID 28813030
- [Background] Xie B, Unger JB, Gallaher P, Johnson CA, Wu Q, Chou CP. Overweight, body image, and depression in Asian and Hispanic adolescents. Am J Health Behav. 2010 Jul-Aug;34(4):476-88. doi: 10.5993/ajhb.34.4.9. PMID 20218759
- [Background] McGuire MT, Wing RR, Klem ML, Lang W, Hill JO. What predicts weight regain in a group of successful weight losers? J Consult Clin Psychol. 1999 Apr;67(2):177-85. doi: 10.1037//0022-006x.67.2.177. PMID 10224727
- [Background] Sarwer DB, von Sydow Green A, Vetter ML, Wadden TA. Behavior therapy for obesity: where are we now? Curr Opin Endocrinol Diabetes Obes. 2009 Oct;16(5):347-52. doi: 10.1097/MED.0b013e32832f5a79. PMID 19623061
- [Background] Blomain ES, Dirhan DA, Valentino MA, Kim GW, Waldman SA. Mechanisms of Weight Regain following Weight Loss. ISRN Obes. 2013 Apr 16;2013:210524. doi: 10.1155/2013/210524. eCollection 2013. PMID 24533218
- [Background] de Jonge L, Bray GA, Smith SR, Ryan DH, de Souza RJ, Loria CM, Champagne CM, Williamson DA, Sacks FM. Effect of diet composition and weight loss on resting energy expenditure in the POUNDS LOST study. Obesity (Silver Spring). 2012 Dec;20(12):2384-9. doi: 10.1038/oby.2012.127. Epub 2012 May 7. PMID 22627912
- [Background] Ebbeling CB, Swain JF, Feldman HA, Wong WW, Hachey DL, Garcia-Lago E, Ludwig DS. Effects of dietary composition on energy expenditure during weight-loss maintenance. JAMA. 2012 Jun 27;307(24):2627-34. doi: 10.1001/jama.2012.6607. PMID 22735432
- [Background] Larsen TM, Dalskov SM, van Baak M, Jebb SA, Papadaki A, Pfeiffer AF, Martinez JA, Handjieva-Darlenska T, Kunesova M, Pihlsgard M, Stender S, Holst C, Saris WH, Astrup A; Diet, Obesity, and Genes (Diogenes) Project. Diets with high or low protein content and glycemic index for weight-loss maintenance. N Engl J Med. 2010 Nov 25;363(22):2102-13. doi: 10.1056/NEJMoa1007137. PMID 21105792
- [Background] Montesi L, El Ghoch M, Brodosi L, Calugi S, Marchesini G, Dalle Grave R. Long-term weight loss maintenance for obesity: a multidisciplinary approach. Diabetes Metab Syndr Obes. 2016 Feb 26;9:37-46. doi: 10.2147/DMSO.S89836. eCollection 2016. PMID 27013897
- [Background] DiBonaventura Md, Chapman GB. The effect of barrier underestimation on weight management and exercise change. Psychol Health Med. 2008 Jan;13(1):111-22. doi: 10.1080/13548500701426711. PMID 18066924
- [Background] Brown SP, Eason JM, Miller WC. Ergometer and calorimetry: the measurement of work and energy. In: Brown SP, Eason JM, Miller WC. Exercise physiology: basis of human movement in health and disease. Philadelphia: Lippincott Williams & Wilkins; 2006.
- [Background] Plowman SA, Smith DL. Aerobic metabolism during exercise. In: Plowman SA, Smith DL. Exercise physiology for health, fitness, and performance. 4th ed. Philadelphia: Lippincott Williams & Wilkins; 2014.
- [Background] Manore MM, Meyer N, Thompson JL. Energy and nutrient balance. In: Manore MM, Meyer N, Thompson JL. Sport nutrition for health and performance. 2nd ed. Illinois: Human Kinetics; 2009.
- [Background] Valtuena S, Salas-Salvado J, Lorda PG. The respiratory quotient as a prognostic factor in weight-loss rebound. Int J Obes Relat Metab Disord. 1997 Sep;21(9):811-7. doi: 10.1038/sj.ijo.0800480. PMID 9376895
- [Background] Kanaley JA, Weatherup-Dentes MM, Alvarado CR, Whitehead G. Substrate oxidation during acute exercise and with exercise training in lean and obese women. Eur J Appl Physiol. 2001 Jul;85(1-2):68-73. doi: 10.1007/s004210100404. PMID 11513323
- [Background] Frayn KN. Calculation of substrate oxidation rates in vivo from gaseous exchange. J Appl Physiol Respir Environ Exerc Physiol. 1983 Aug;55(2):628-34. doi: 10.1152/jappl.1983.55.2.628. PMID 6618956
- [Background] Katzmarzyk PT, Perusse L, Tremblay A, Bouchard C. No association between resting metabolic rate or respiratory exchange ratio and subsequent changes in body mass and fatness: 5-1/2 year follow-up of the Quebec family study. Eur J Clin Nutr. 2000 Aug;54(8):610-4. doi: 10.1038/sj.ejcn.1601053. PMID 10951508
- [Background] Marion-Latard F, Crampes F, Zakaroff-Girard A, De Glisezinski I, Harant I, Stich V, Thalamas C, Riviere D, Lafontan M, Berlan M. Post-exercise increase of lipid oxidation after a moderate exercise bout in untrained healthy obese men. Horm Metab Res. 2003 Feb;35(2):97-103. doi: 10.1055/s-2003-39051. PMID 12734789
- [Background] van Aggel-Leijssen DP, Saris WH, Wagenmakers AJ, Hul GB, van Baak MA. The effect of low-intensity exercise training on fat metabolism of obese women. Obes Res. 2001 Feb;9(2):86-96. doi: 10.1038/oby.2001.11. PMID 11316351
- [Background] Helge JW, Fraser AM, Kriketos AD, Jenkins AB, Calvert GD, Ayre KJ, Storlien LH. Interrelationships between muscle fibre type, substrate oxidation and body fat. Int J Obes Relat Metab Disord. 1999 Sep;23(9):986-91. doi: 10.1038/sj.ijo.0801030. PMID 10490806
- [Background] Crisp NA, Guelfi KJ, Braham R, Licari M. Substrate oxidation in overweight boys at rest, during exercise and acute post-exercise recovery. Int J Pediatr Obes. 2011 Jun;6(2-2):e615-21. doi: 10.3109/17477166.2010.543684. Epub 2011 Jan 18. PMID 21244226
- [Background] Lanzi S, Codecasa F, Cornacchia M, Maestrini S, Salvadori A, Brunani A, Malatesta D. Fat oxidation, hormonal and plasma metabolite kinetics during a submaximal incremental test in lean and obese adults. PLoS One. 2014 Feb 11;9(2):e88707. doi: 10.1371/journal.pone.0088707. eCollection 2014. PMID 24523934
- [Background] Rosenkilde M, Nordby P, Nielsen LB, Stallknecht BM, Helge JW. Fat oxidation at rest predicts peak fat oxidation during exercise and metabolic phenotype in overweight men. Int J Obes (Lond). 2010 May;34(5):871-7. doi: 10.1038/ijo.2010.11. Epub 2010 Feb 16. PMID 20157319
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Sakaguchi T, Arase K, Bray GA. Sympathetic activity and food intake of rats with ventromedial hypothalamic lesions. Int J Obes. 1988;12(4):285-91. PMID 3198309
- [Background] Yoshida T, Kemnitz JW, Bray GA. Lateral hypothalamic lesions and norepinephrine turnover in rats. J Clin Invest. 1983 Sep;72(3):919-27. doi: 10.1172/JCI111063. PMID 6886011
- [Background] Bray GA. Obesity--a disease of nutrient or energy balance? Nutr Rev. 1987 Feb;45(2):33-43. doi: 10.1111/j.1753-4887.1987.tb07437.x. No abstract available. PMID 3550538
- [Background] Guarino D, Nannipieri M, Iervasi G, Taddei S, Bruno RM. The Role of the Autonomic Nervous System in the Pathophysiology of Obesity. Front Physiol. 2017 Sep 14;8:665. doi: 10.3389/fphys.2017.00665. eCollection 2017. PMID 28966594
- [Background] Goldfield GS, Kenny GP, Alberga AS, Prud'homme D, Hadjiyannakis S, Gougeon R, Phillips P, Tulloch H, Malcolm J, Doucette S, Wells GA, Ma J, Cameron JD, Sigal RJ. Effects of aerobic training, resistance training, or both on psychological health in adolescents with obesity: The HEARTY randomized controlled trial. J Consult Clin Psychol. 2015 Dec;83(6):1123-35. doi: 10.1037/ccp0000038. Epub 2015 Aug 31. PMID 26322787
- [Background] Baruth M, Sharpe PA, Parra-Medina D, Wilcox S. Perceived barriers to exercise and healthy eating among women from disadvantaged neighborhoods: results from a focus groups assessment. Women Health. 2014;54(4):336-53. doi: 10.1080/03630242.2014.896443. PMID 24617795
- [Background] Draper CE, Davidowitz KJ, Goedecke JH. Perceptions relating to body size, weight loss and weight-loss interventions in black South African women: a qualitative study. Public Health Nutr. 2016 Feb;19(3):548-56. doi: 10.1017/S1368980015001688. Epub 2015 May 26. PMID 26006784
- [Background] Blow JA, Taylor T, Cooper TV, Redfearn CK. Correlates of weight concern and control in a Hispanic college student sample. Eat Behav. 2010 Jan;11(1):6-10. doi: 10.1016/j.eatbeh.2009.08.001. Epub 2009 Aug 18. PMID 19962114
- [Background] Martins C, Kazakova I, Ludviksen M, Mehus I, Wisloff U, Kulseng B, Morgan L, King N. High-Intensity Interval Training and Isocaloric Moderate-Intensity Continuous Training Result in Similar Improvements in Body Composition and Fitness in Obese Individuals. Int J Sport Nutr Exerc Metab. 2016 Jun;26(3):197-204. doi: 10.1123/ijsnem.2015-0078. Epub 2015 Oct 19. PMID 26479856
- [Background] Pillard F, Moro C, Harant I, Garrigue E, Lafontan M, Berlan M, Crampes F, de Glisezinski I, Riviere D. Lipid oxidation according to intensity and exercise duration in overweight men and women. Obesity (Silver Spring). 2007 Sep;15(9):2256-62. doi: 10.1038/oby.2007.268. PMID 17890494
- [Background] Layden JD, Patterson MJ, Nimmo MA. Effects of reduced ambient temperature on fat utilization during submaximal exercise. Med Sci Sports Exerc. 2002 May;34(5):774-9. doi: 10.1097/00005768-200205000-00008. PMID 11984294
- [Background] Zumoff B, Strain GW, Miller LK, Rosner W. Twenty-four-hour mean plasma testosterone concentration declines with age in normal premenopausal women. J Clin Endocrinol Metab. 1995 Apr;80(4):1429-30. doi: 10.1210/jcem.80.4.7714119.
- [Background] Wu YT, Nielsen DH, Cassady SL, Cook JS, Janz KF, Hansen JR. Cross-validation of bioelectrical impedance analysis of body composition in children and adolescents. Phys Ther. 1993 May;73(5):320-8. doi: 10.1093/ptj/73.5.320. PMID 8469716
- [Background] Lukaski HC, Bolonchuk WW, Hall CB, Siders WA. Validation of tetrapolar bioelectrical impedance method to assess human body composition. J Appl Physiol (1985). 1986 Apr;60(4):1327-32. doi: 10.1152/jappl.1986.60.4.1327. PMID 3700310
- [Background] Segal KR, Van Loan M, Fitzgerald PI, Hodgdon JA, Van Itallie TB. Lean body mass estimation by bioelectrical impedance analysis: a four-site cross-validation study. Am J Clin Nutr. 1988 Jan;47(1):7-14. doi: 10.1093/ajcn/47.1.7. PMID 3337041
- [Background] Jackson AS, Pollock ML, Graves JE, Mahar MT. Reliability and validity of bioelectrical impedance in determining body composition. J Appl Physiol (1985). 1988 Feb;64(2):529-34. doi: 10.1152/jappl.1988.64.2.529. PMID 3372410
- [Background] Sanchez-Miguel PA, Gonzalez JJP, Sanchez-Oliva D, Alonso DA, Leo FM. The importance of body satisfaction to physical self-concept and body mass index in Spanish adolescents. Int J Psychol. 2019 Aug;54(4):521-529. doi: 10.1002/ijop.12488. Epub 2018 Apr 6. PMID 29633263
- [Background] Thompson JK, Altabe MN. Psychometric qualities of the Figure Rating Scale. Int J Eat Disord. 1991;10:615-9.
- [Background] Cash TF. The Multidimensional Body-Self Relations Questionnaire. MBRSQ Users' Manual (Third Revision). 2000.
- [Background] Sallis JF, Haskell WL, Wood PD, Fortmann SP, Rogers T, Blair SN, Paffenbarger RS Jr. Physical activity assessment methodology in the Five-City Project. Am J Epidemiol. 1985 Jan;121(1):91-106. doi: 10.1093/oxfordjournals.aje.a113987. PMID 3964995
- [Background] Lee YS, Chu CY, Lin KF. Application of Physical Activity Scales/Questionnaires in Taiwan. J Exerc Physiol Fit. 2010;11:1-12.
- [Background] Dishman RK, Steinhardt M. Reliability and concurrent validity for a 7-d re-call of physical activity in college students. Med Sci Sports Exerc. 1988 Feb;20(1):14-25. doi: 10.1249/00005768-198802000-00003. PMID 3343912
- [Background] Karlsson J, Persson LO, Sjostrom L, Sullivan M. Psychometric properties and factor structure of the Three-Factor Eating Questionnaire (TFEQ) in obese men and women. Results from the Swedish Obese Subjects (SOS) study. Int J Obes Relat Metab Disord. 2000 Dec;24(12):1715-25. doi: 10.1038/sj.ijo.0801442. PMID 11126230
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Bohrer BK, Forbush KT, Hunt TK. Are common measures of dietary restraint and disinhibited eating reliable and valid in obese persons? Appetite. 2015 Apr;87:344-51. doi: 10.1016/j.appet.2014.12.226. Epub 2015 Jan 9. PMID 25582416
- [Background] Maust D, Cristancho M, Gray L, Rushing S, Tjoa C, Thase ME. Psychiatric rating scales. Handb Clin Neurol. 2012;106:227-37. doi: 10.1016/B978-0-444-52002-9.00013-9. No abstract available. PMID 22608624
- [Background] Paiva-Medeiros PF, Duarte-Guerra LS, Santo MA, Lotufo-Neto F, Wang YP. Psychometric Properties of the Montgomery-Asberg Depression Rating Scale in Severely Obese Patients. Span J Psychol. 2015 Sep 14;18:E69. doi: 10.1017/sjp.2015.072. PMID 26364907
- [Background] Schaefer LM, Harriger JA, Heinberg LJ, Soderberg T, Kevin Thompson J. Development and validation of the sociocultural attitudes towards appearance questionnaire-4-revised (SATAQ-4R). Int J Eat Disord. 2017 Feb;50(2):104-117. doi: 10.1002/eat.22590. Epub 2016 Aug 19. PMID 27539814
- [Background] Rosen JC, Jones A, Ramirez E, Waxman S. Body Shape Questionnaire: studies of validity and reliability. Int J Eat Disord. 1996 Nov;20(3):315-9. doi: 10.1002/(SICI)1098-108X(199611)20:33.0.CO;2-Z. PMID 8912044